CLINICAL TRIAL: NCT03449797
Title: The Intra-Procedural Cortisol Assay During Adrenal Vein Sampling: Rationale andDesign of A Randomized Study (I-PADUA)
Brief Title: Rapid Cortisol Assay in Adrenal Vein Sampling
Acronym: I-PADUA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Padova (Other)
Responsible Party: Principal Investigator, Gian Paolo Rossi, MD, FAHA, FACC, Professor of Medicine, University Hospital Padova
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: UHPadova
Record Dates: First submitted 2018-02-22; First posted 2018-02-28 (Actual); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Primary Aldosteronism Due to Aldosterone Producing Adenoma
Keywords: aldosterone; cortisol; adrenal vein sampling; primary aldosteronism
MeSH Terms: conditions — Hyperaldosteronism

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Sham Comparator): AAVS performed with no intraprocedural rapid cortisol assay
  Interventions: Procedure: AVS performed with no intraprocedural rapid cortisol assay
- Group B (Experimental): AVS performed plus intraprocedural rapid cortisol assay
  Interventions: Procedure: AVS performed plus intraprocedural rapid cortisol assay

INTERVENTIONS:
Procedure: AVS performed with no intraprocedural rapid cortisol assay — AVS performed plus intraprocedural rapid cortisol assay
  Arms: Group A
Procedure: AVS performed plus intraprocedural rapid cortisol assay — Adrenal vein sampling performed according to usual clinical practice without intraprocedural rapid cortisol assay
  Arms: Group B

SUMMARY:
Background: Adrenal vein sampling (AVS) is the gold standard test for the subtyping of primary aldosteronism (PA). This procedure is hampered by unsuccessful bilateral cannulation of adrenal veins, which can occur in up to two thirds of the cases depending on the cutoff of the selectivity index used. The rapid intra-procedural cortisol assay (IRCA) can increase the rate of bilateral success of AVS. This can be proven using a randomized prospective study design approach.

Aim: We will therefore evaluate if an IRCA-guided AVS strategy can increase the rate of selectivity and thus the success rate of adrenal vein catheterization.

Methods: Consecutive patients with a biochemical diagnosis of PA, seeking surgical cure, will be randomized to undergo AVS according to an IRCA-sham or an IRCA-guided procedure.

Experimental and endpoint will be the rate of bilaterally selective AVS studies as defined by a selective index cutoff > 2.00 value under baseline (unstimulated) conditions. With 100 patients submitted to AVS with a normal procedure and 100 patients undergoing AVS with IRCA, it has been estimated that the study has 82% power to detect a significant difference of 18% at a two-sided 0.05 significance level between arms.

Expected results. Given this power we expect to the able to determine if IRCA is useful or not for improving the success rate of AVS. Given the current disastrous situation regarding the clinical use of AVS this will be a major accomplishment in the field of the subtyping of PA.

DETAILED DESCRIPTION:
Primary aldosteronism (PA) is a common form of hypertension caused by excess aldosterone secretion: it involves over 11% of the patients referred to specialized hypertension centres [1], about one fifth of those with drug-resistant hypertension [2] and about 6% of the hypertensive patients seen in general practice [3].

PA is held to cause cardiovascular disease in excess of the degree of blood pressure elevation, which translates into a high rate of cardiovascular events. These ominous consequences can be prevented with a timely diagnosis. Once the diagnosis of PA has been made, the decision to proceed further with surgical or medical treatment depends on identification of the PA subtype. In fact, adrenalectomy, can be necessary in up to two thirds of the PA cases [1], and was shown to regress cardiovascular damage and prevent CV events at long-term [4]. Therefore, identification of PA followed by subtyping entails fundamental steps that can be particularly beneficial in some subgroups of patients as those with drug-resistant hypertension, who are at high cardiovascular risk of PA [2].

Adrenalectomy is indicated only once a lateralized aldosterone excess has been identified by adrenal vein sampling (AVS). This is a technically challenging procedure because placing the catheter's tip within the tiny and short right adrenal vein is difficult. Samples are, therefore, often obtained from at or near the orifice of the vein, which can lead to dilution of the adrenal hormones, and thus to non selective studies. Unfortunately, accomplishment bilateral selectivity was disappointingly low, particularly if high cutoff values of the selectivity index are used, as shown by the largest study ever performed worldwide. To overcome this limitation several methods have recently been proposed, including stimulation with cosyntropin or metoclopramide [5-10], use of alternative biomarkers, as for example, plasma metanephrines or androstenedione that have a step-up between adrenal vein and inferior vena cava (IVC) higher than cortisol [11], and the intra-procedural rapid cortisol assay (IRCA). The latter can improve the success rate of AVS, particularly at a stage when radiologists are gaining experience with the procedure. Accordingly, several centres have adopted this practice after its introduction [12] and reported anecdotal successes, but logistic problems have prevented widespread use of IRCA in clinical practice [13].

Recently a kit for the semi-quantitative IRCA has been developed [14], which lends itself to routine clinical use owing to its simplicity, ease, and speed of use. Yet, the advantages of exploiting an IRCA-based strategy for improving the success rate in achieving selectivity of AVS has been proven only in one randomized clinical trial (RCT) carried out in Japan, which involved 7 centres, most of which had no or, a limited experience with AVS [14].

RTCs represent the basis for evidence-based and high-grade class of recommendations in practice guidelines. Therefore, we plan to test the hypothesis that the IRCA during AVS could improve the rate of bilaterally selective AVS studies over that accomplished by a routine AVS protocol even when used at referral centres that routinely perform this diagnostic procedure.

Methods Consecutive patients with biochemical diagnosis of PA seeking surgical cure of PA will be recruited for this study, according to current guidelines [15]. These patients have a compelling indication to AVS before being referred or not for adrenalectomy [9]. The only exclusion criteria will be: a) refusal of the centre to participate in the study; b) refusal of the patient to undergo AVS , c) contraindications to the general anaesthesia that is required for laparoscopic adrenalectomy; d) cortisol co-secreting adenoma. The latter criterion is necessary because, given the cortisol-derived selectivity index (see below) primary endpoint chosen, inclusion of these tumours would introduce an obvious confounding bias on results [16].

Study design The outlay of this prospective randomized two-arm multicentre study, and its primary endpoint are summarized below. Randomization will be performed with a specific algorithm as provided in a the SPSSS statistical package. The study will last until 220 patients will be recruited and randomly assigned to either arm considering the possibility of a 10% dropout rate. Data collection will be performed by means of a specific form created ad hoc for the AVIS Study and modified as required [17]. The assignment to either arm will be coded and the data analysis for the primary end-point will be performed by investigators blindly to arm assignment.

In the IRCA arm, the plasma obtained simultaneously from each adrenal vein and the IVC will be tested with typical cortisol assay and in case of non selective results catheters will be repositioned until selective results will be obtained until a maximum of 3 attempts. In the IRCA-sham group only the IVC plasma will be tested and no catheter's repositioning will be undertaken.

The AVS will be performed according to the protocol recently described with bilaterally simultaneous sampling but without metoclopramide stimulation [5]. The IRCA will be performed using the procedure on-going at each participating centre. This implies using either an in-house made, or the commercially available semi-quantitative kit (Trust Medical Support Co., Ltd. Fukuoka, Japan).

All procedures will be according to good clinical practice and to the Declaration of Helsinki and the study will started after approval of the Ethics Committee of the University of Padua and, if necessary, of the participating centres.

Primary endpoint Selectivity will be determined on both side by using a value of the selectivity index > 2.00 as defined in an Expert Consensus Statement of AVS [9]. The definition of the selectivity index (SI) has been already reported [16]; briefly, this is the ratio between plasma cortisol concentration in each adrenal vein and in the infrarenal inferior vena cava blood. The selectivity index will be determined based on measurement of cortisol in the central laboratory of each center. For quality control purposes aliquots of plasma will be collected in heparina and EDTA for metanephrine and androstenedione measurement in the core lab of the coordinating center.

Sample size calculation and statistical analysis We have calculated that with 100 patients submitted to AVS with a normal procedure (Group A) and 100 patients undergoing AVS with IRCA (Group B), the study will have a 82% power of detecting a significant difference of 18% at a two-sided 0.05 significance level, assuming that the SI in Group A is 67% and in Group B is 85 %.

Discussion Currently randomized clinical trials entail the best methodology to provide high-grade class of recommendation and high level of evidence. Therefore, they represent an inevitable step for introducing novel diagnostic and therapeutic strategies where uncertainties still exist as the subtyping of PA by means of adrenal vein sampling.

In fact, the recent publication of SPARTACUS, a randomized clinical trial in the field of a subtyping of PA, has challenged the Endocrine Society Practice guidelines recommendation of performing AVS in all patients seeking surgical cure of PA, who are reasonable candidate for adrenalectomy in general anaesthesia,according to guidelines. In fact, it showed no outcome differences between an AVS- and a computed tomography- based strategy for PA subtyping [18], thus adding a good deal of fuel to the controversy on whether to submit or not all PA to AVS before referring them for adrenalectomy. Although the study was widely criticized and, moreover was not adequately powered, it is altogether evident that in current clinical practice the diagnostic performance of AVS is far from optimal worldwide as shown in the AVIS Study.

Hence, efforts aimed at proving the usefulness of novel strategies for improving the rate of selective AVS studies entail a much worth effort, which should be undertaken by exploiting the RCT methodology. We therefore expect that studies, as the one herein described, being adequately powered from the statistical standpoint, can provide a definitive answer to the question of the whether IRCA can increase the rate of selectivity of AVS. Specifically, we expect to be able to detect a difference of about 18%, e.g. from 67% to 85%, in the rate of bilateral selectivity between the arms.

To date, only one study using a single commercially available kit for semiquantitative IRCA has exploited use of a randomized design to prove the usefulness of this strategy for improving the success rate of AVS in Japan [14]. Unfortunately, most recruited centres and radiologists were not proficient in performing the procedure, which might explain the remarkable advantage seen with IRCA. Hence, it remains to be demonstrated if use of the IRCA can provide similar advantages in different settings as referral centres endowed with radiologists that are proficient in performing AVS. Once verified, or disproved, this hypothesis will have an impact on widespread adoption or abandoning of the IRCA in clinical practice.

In summary, testing the usefulness of an IRCA for increasing the success rate of AVS in a multi-centre randomized clinical trial as that herein described is expected to fill an important gap of information in the field of subtyping of PA. This increased knowledge will ultimately improve the diagnostic use of AVS, which remain the key test for referring PA patients for adrenalectomy.

ELIGIBILITY:
Inclusion Criteria: According to current guidelines consecutive patients with biochemical diagnosis of PA, who seek surgical cure of PA will be recruited for this study.These patients have a compelling indication to AVS before being referred or not for adrenalectomy.

-

Exclusion Criteria: i) refusal of the center's to participate in the study; ii)refusal of the patientto undergo AVS and/or contraindications to the general anesthesia that is required for laparoscopic adrenalectomy; iii) cortisol -and aldosterone co-secreting adenoma.

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of selectivity of the sample | two years
  Selectivity will be determined on both side by using a value of the selectivity index > 2.00 as defined in an Expert Consensus Statement of AVS. Selectivity is the ratio between plasma cortisol concentration in each adrenal vein and in the infrarenal inferior vena cava blood.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rossi GP, Bernini G, Caliumi C, Desideri G, Fabris B, Ferri C, Ganzaroli C, Giacchetti G, Letizia C, Maccario M, Mallamaci F, Mannelli M, Mattarello MJ, Moretti A, Palumbo G, Parenti G, Porteri E, Semplicini A, Rizzoni D, Rossi E, Boscaro M, Pessina AC, Mantero F; PAPY Study Investigators. A prospective study of the prevalence of primary aldosteronism in 1,125 hypertensive patients. J Am Coll Cardiol. 2006 Dec 5;48(11):2293-300. doi: 10.1016/j.jacc.2006.07.059. Epub 2006 Nov 13. PMID 17161262
- [Result] Douma S, Petidis K, Doumas M, Papaefthimiou P, Triantafyllou A, Kartali N, Papadopoulos N, Vogiatzis K, Zamboulis C. Prevalence of primary hyperaldosteronism in resistant hypertension: a retrospective observational study. Lancet. 2008 Jun 7;371(9628):1921-6. doi: 10.1016/S0140-6736(08)60834-X. PMID 18539224
- [Result] Olivieri O, Ciacciarelli A, Signorelli D, Pizzolo F, Guarini P, Pavan C, Corgnati A, Falcone S, Corrocher R, Micchi A, Cressoni C, Blengio G. Aldosterone to Renin ratio in a primary care setting: the Bussolengo study. J Clin Endocrinol Metab. 2004 Sep;89(9):4221-6. doi: 10.1210/jc.2003-032179. PMID 15356010
- [Result] Rossi GP, Cesari M, Cuspidi C, Maiolino G, Cicala MV, Bisogni V, Mantero F, Pessina AC. Long-term control of arterial hypertension and regression of left ventricular hypertrophy with treatment of primary aldosteronism. Hypertension. 2013 Jul;62(1):62-9. doi: 10.1161/HYPERTENSIONAHA.113.01316. Epub 2013 May 6. PMID 23648698
- [Result] Rossitto G, Miotto D, Battistel M, Barbiero G, Maiolino G, Bisogni V, Sanga V, Rossi GP. Metoclopramide unmasks potentially misleading contralateral suppression in patients undergoing adrenal vein sampling for primary aldosteronism. J Hypertens. 2016 Nov;34(11):2258-65. doi: 10.1097/HJH.0000000000001082. PMID 27512976
- [Result] Weinberger MH, Grim CE, Hollifield JW, Kem DC, Ganguly A, Kramer NJ, Yune HY, Wellman H, Donohue JP. Primary aldosteronism: diagnosis, localization, and treatment. Ann Intern Med. 1979 Mar;90(3):386-95. doi: 10.7326/0003-4819-90-3-386. PMID 218482
- [Result] Young WF Jr, Stanson AW, Grant CS, Thompson GB, van Heerden JA. Primary aldosteronism: adrenal venous sampling. Surgery. 1996 Dec;120(6):913-9; discussion 919-20. PMID 8957473
- [Result] Young WF, Stanson AW, Thompson GB, Grant CS, Farley DR, van Heerden JA. Role for adrenal venous sampling in primary aldosteronism. Surgery. 2004 Dec;136(6):1227-35. doi: 10.1016/j.surg.2004.06.051. PMID 15657580
- [Result] Rossi GP, Auchus RJ, Brown M, Lenders JW, Naruse M, Plouin PF, Satoh F, Young WF Jr. An expert consensus statement on use of adrenal vein sampling for the subtyping of primary aldosteronism. Hypertension. 2014 Jan;63(1):151-60. doi: 10.1161/HYPERTENSIONAHA.113.02097. Epub 2013 Nov 11. PMID 24218436
- [Result] Seccia TM, Miotto D, De Toni R, Pitter G, Mantero F, Pessina AC, Rossi GP. Adrenocorticotropic hormone stimulation during adrenal vein sampling for identifying surgically curable subtypes of primary aldosteronism: comparison of 3 different protocols. Hypertension. 2009 May;53(5):761-6. doi: 10.1161/HYPERTENSIONAHA.108.128553. Epub 2009 Apr 6. PMID 19349554
- [Result] Lenders JW, Duh QY, Eisenhofer G, Gimenez-Roqueplo AP, Grebe SK, Murad MH, Naruse M, Pacak K, Young WF Jr; Endocrine Society. Pheochromocytoma and paraganglioma: an endocrine society clinical practice guideline. J Clin Endocrinol Metab. 2014 Jun;99(6):1915-42. doi: 10.1210/jc.2014-1498. PMID 24893135
- [Result] Woods JJ, Sampson ML, Ruddel ME, Remaley AT. Rapid intraoperative cortisol assay: design and utility for localizing adrenal tumors by venous sampling. Clin Biochem. 2000 Aug;33(6):501-3. doi: 10.1016/s0009-9120(00)00141-7. No abstract available. PMID 11074243
- [Result] Mengozzi G, Rossato D, Bertello C, Garrone C, Milan A, Pagni R, Veglio F, Mulatero P. Rapid cortisol assay during adrenal vein sampling in patients with primary aldosteronism. Clin Chem. 2007 Nov;53(11):1968-71. doi: 10.1373/clinchem.2007.092080. Epub 2007 Sep 27. PMID 17901112
- [Result] Yoneda T, Karashima S, Kometani M, Usukura M, Demura M, Sanada J, Minami T, Koda W, Gabata T, Matsui O, Idegami K, Takamura Y, Tamiya E, Oe M, Nakai M, Mori S, Terayama N, Matsuda Y, Kamemura K, Fujii S, Seta T, Sawamura T, Okuda R, Takeda Y, Hayashi K, Yamagishi M, Takeda Y. Impact of New Quick Gold Nanoparticle-Based Cortisol Assay During Adrenal Vein Sampling for Primary Aldosteronism. J Clin Endocrinol Metab. 2016 Jun;101(6):2554-61. doi: 10.1210/jc.2016-1011. Epub 2016 Mar 24. PMID 27011114
- [Result] Funder JW, Carey RM, Mantero F, Murad MH, Reincke M, Shibata H, Stowasser M, Young WF Jr. The Management of Primary Aldosteronism: Case Detection, Diagnosis, and Treatment: An Endocrine Society Clinical Practice Guideline. J Clin Endocrinol Metab. 2016 May;101(5):1889-916. doi: 10.1210/jc.2015-4061. Epub 2016 Mar 2. PMID 26934393
- [Result] Rossi GP, Ganzaroli C, Miotto D, De Toni R, Palumbo G, Feltrin GP, Mantero F, Pessina AC. Dynamic testing with high-dose adrenocorticotrophic hormone does not improve lateralization of aldosterone oversecretion in primary aldosteronism patients. J Hypertens. 2006 Feb;24(2):371-9. doi: 10.1097/01.hjh.0000202818.10459.96. PMID 16508586